CLINICAL TRIAL: NCT06257355
Title: A Two-Arm Open-Label Study to Evaluate the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Subjects With Corneal Scars
Brief Title: Study to Evaluate the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Subjects With Corneal Scars
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Claris Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSB-C23-002
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Corneal Scar
MeSH Terms: conditions — Corneal Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSB-001 QID (Experimental): One drop CSB-001 four times daily for 14 days in the study eye
  Interventions: Biological: CSB-001 Ophthalmic Solution 0.1%
- CSB-001 TID (Experimental): One drop CSB-001 three times daily for 14 days in the study eye
  Interventions: Biological: CSB-001 Ophthalmic Solution 0.1%

INTERVENTIONS:
Biological: CSB-001 Ophthalmic Solution 0.1% — CSB-001: human recombinant dHGF (5-amino acid deleted hepatocyte growth factor)

SUMMARY:
This study will enroll subjects with recently formed corneal scars that resulted from a corneal insult presenting and diagnosed within the past approximately 30 days and not less than approximately 7 days. All subjects will be assigned to CSB-001 investigational treatment on Day 1. All subjects will dose with CSB-001 four times daily or three times daily starting on Day 1 and continue until Day 14. Subjects with a resolved scar at Day 7 will discontinue dosing and return to the clinic on Day 14. Subjects will return on Days 21, 28, 56, and Month 3 for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Centrally or paracentrally located scar approximately ≤5 mm and ≥2 mm in the greatest diameter and with a portion of the scar within approximately 3.5 mm of the optical center of the cornea assessed at Screening and confirmed at Baseline, and subject reports ability to detect any effect of scar on any element of vision.
* Eye with a recent corneal insult approximately ≤30 days and ≥7 days from the Screening Visit.
* Corneal insult includes but is not limited to mechanical / chemical / thermal injury, bacterial keratitis, PRK, and contact lens related ulcer.
* Eye with observed rate of epithelialization that in the investigator's opinion does not demonstrate clinical characteristics of a slow healing (persistent defect) cornea.
* Subjects must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

* Corneal scar that encompasses more than approximately 50% of the depth of the remaining stroma as guided by ASOCT image at the Screening Visit.
* Maximum scar diameter greater than approximately 5 mm without prior approval by the Sponsor based on Screening Visit images.
* No portion of the scar is within the approximate 3.5 mm of the optical center of the cornea based on Screening Visit images.
* Any active ocular infection in the opinion of the investigator (bacterial, viral, fungal, or protozoal) at the Screening or Day 1 Visits. Subjects with an active bacterial infection at the Screening or Day 1 Visit in the opinion of the investigator may be rescheduled to reassess the status of the infection and continue in the study if infection is deemed not active.
* Ocular surgery planned during the study treatment period.
* Presence or history of any ocular or systemic disorder, condition or procedure that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct.

Note: Other inclusion/exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety as Assessed by Adverse Event Reporting | Day 1 through Day 56
  Incidence of ocular and systemic adverse events
Safety as Assessed by Slit-lamp Biomicroscopy | Screening through Day 56
  Change from baseline in staining using NEI scale (0 = absent to 3 = severe for 5 areas of the cornea) with Grade 0 (no staining) to maximum of Grade 15
Safety as Assessed by Best-Corrected Distance Visual Acuity | Screening through Day 56
  Change from baseline using the Early Treatment Diabetic Retinopathy Study (EDTRS) visual acuity chart

SECONDARY OUTCOMES:
Efficacy as Assessed by Area of Corneal Scar | Screening through Day 56
  Area of corneal scar as measured by slit lamp and anterior segment optical coherence tomography (AS-OCT) imaging
Efficacy as Assessed by Maximum Depth of Cornea Scar | Screening through Day 56
  Depth measured with AS-OCT imaging
Efficacy as Assessed by Volume of Scar | Screening through Day 56
  Volume measured with AS-OCT imaging
Efficacy as Assessed by Density of Scar | Screening through Day 56
  Density based on AS-OCT and Pentacam imaging
Efficacy as Assessed by Contrast Sensitivity | Screening through Day 56
  Contrast sensitivity measured using Pelli-Robson chart
Efficacy as Assessed by Distance Visual Acuity | Screening through Day 56
  Visual acuity measured using the EDTRS visual acuity chart

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Loma Linda University Eye Institute, Loma Linda, California
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Francis Price Jr, MD, Indianapolis, Indiana
  - Minnesota Eye Consultants, Minnetonka, Minnesota
  - Legacy Devers Eye Institute, Portland, Oregon
  - Stuart A. Terry, MD PA, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No